CLINICAL TRIAL: NCT00221520
Title: Trial on The Efficacy of Sedation in Mechanically Ventilated Critically Ill Patients
Brief Title: Sedation in the Intensive Care Unit
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Geneva (Other)
Collaborators: Swiss National Science Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3200-068312; 2002DR2266
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2007-01

CONDITIONS: Critical Illness; Respiratory Failure
Keywords: Sedation, mechanical ventilation
MeSH Terms: conditions — Critical Illness; Respiratory Insufficiency | interventions — Midazolam

INTERVENTIONS:
Drug: midazolam with 2 different levels of sedation scores

SUMMARY:
High-risk critically ill patients often require mechanical ventilation either to primarily support the respiratory function or when the ventilation is insufficient to maintain adequate gas exchanges as a result of other organ impairment. In order to tolerate this aggressive mechanical support, enhance patient synchrony with the ventilator, and relieve pain and anxiety, analgesia and sedation are provided. It is suggested that an inappropriate use of sedation and analgesia may prolong the duration of mechanical ventilation and increase the risk of specific adverse outcomes such as ventilator associated pneumonia. Despite the widespread use of sedation, little information is available concerning the effect of varying the level of sedation on patients' subsequent mental health. We designed a randomized controlled trial to investigate the efficacy of sedation with the goal of maintaining the patient cooperative and interactive compared to the administration of sedation with the goal of maintaining the patient sedated. The first goal will be achieved by a discontinuous injection of a sedative, while the second goal will be achieved by a continuous infusion of the same sedative. In both groups pain relief will be provided in the same fashion with equal endpoints on a pain scoring scale. Our primary aim is to investigate whether differences in the occurrence of post-traumatic stress disorders (PTSD), anxiety, and depression are related to the choice of sedation-analgesia strategies. Secondary endpoints include the length of ICU stay, as indicated by the time to discharge from the ICU, the time to separation from mechanical ventilation, the rates of pulmonary and extra-pulmonary complications, and hospital length of stay. These endpoints will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients requiring mechanical ventilation

Exclusion Criteria:

* Neurological conditions or neuromuscular disease
* Chronic renal failure, liver failure
* Allergy to benzodiazepines or morphine
* Drug overdose
* Pregnancy
* Non-cooperative
* Treatment with HIV protease inhibitors or erythromycin
* Refusal of consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126
Dates: Start 2003-02; Study Completion 2007-01

PRIMARY OUTCOMES:
Post-traumatic stress disorders (PTSD)
Anxiety
Depression

SECONDARY OUTCOMES:
Time to discharge from the Intensive Care Unit
Time to separation from mechanical ventilation
Rates of pulmonary and extra-pulmonary complications Hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Miriam M Treggiari, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland